CLINICAL TRIAL: NCT02796911
Title: Effectiveness of Bovine Derived Xenograft Versus Bioactive Glass With Periodontally Accelerated Osteogenic Orthodontics in Adults
Brief Title: Comparative Study of Different Bone Grafts in Accelerating Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maha A. Bahammam, Associate Professor and Consultant of Periodontology, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 029-16
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Orthodontics
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Corticotomy alone (No Intervention): Group I will be treated with a modified technique of corticotomy assisted orthodontic treatment (CAOT) alone
- Corticotomy + xenograft (Experimental): group II (included 6 females and 5 males) that treated with CAOT combined with bovine derived xenograft (Biogen, Biotecksrl Fermi, Arcugraro VI, Italy);
  Interventions: Drug: Xenograft
- Corticotomy + bioactive glass (Experimental): group III (included 7 females and 4 males) that treated with CAOT combined with bioactive glass (Bio-Glass, Excellence Pharm Inc., Egypt).
  Interventions: Drug: Bioactive glass

INTERVENTIONS:
Drug: Xenograft — group II will be treated with CAOT combined with bovine derived xenograft (Biogen, Biotecksrl Fermi, Arcugraro VI, Italy);
  Other Names: bovine derived xenograft
  Arms: Corticotomy + xenograft
Drug: Bioactive glass — group III will be treated with CAOT combined with bioactive glass (Bio-Glass, Excellence Pharm Inc., Egypt).
  Arms: Corticotomy + bioactive glass

SUMMARY:
Objective: Periodontally accelerated osteogenic orthodontics(PAOO) will minimize treatment time. The current study will be carried to evaluate the effectiveness of different bone grafts with a modified, less invasive corticotomy technique in the treatment of adult patients with moderate crowding.

Subjects and Methods: Thirty orthodontic patients will be selected. Patients were randomly classified into three groups. Group I will be treated with a modified technique of corticotomy, whereas group II will be treated with the same technique combined with PAOO using bovine derived xenograft, and group III will be treated with the same technique combined with PAOO using with bioactive glass. The total duration of active orthodontic treatment will be estimated. Probing depth, bone density and root length will be also evaluated. The measurements will be recorded.

DETAILED DESCRIPTION:
Objective: Periodontally accelerated osteogenic orthodontics(PAOO) combines periodontal therapy with orthodontic therapy, which will minimize treatment time. The current study will be carried to evaluate the effectiveness of bovine derived xenograft versus bioactive glass with a modified, less invasive corticotomy technique in the treatment of adult patients with moderate crowding.

Subjects and Methods: Thirty orthodontic patients will be selected. Patients were randomly classified into three groups. Group I will be treated with a modified technique of corticotomy on the labial side only, whereas group II will be treated with the same technique combined with PAOO using bovine derived xenograft, and group III will be treated with the same technique combined with PAOO using with bioactive glass. The total duration of active orthodontic treatment will be estimated from the time of starting the active orthodontic treatment, immediately following the corticotomy procedure, to the time of debonding. Probing depth will be evaluated clinically whereas bone density and root length will be evaluated radiographically. The measurements will be recorded at day of surgery (baseline) (T1), post-treatment at time of debonding (T2), and 9 months post-treatment (T3).

ELIGIBILITY:
Inclusion Criteria:

* A moderate 4-5mm crowding of the lower anterior teeth
* Good oral hygiene
* Healthy systemic condition

Exclusion Criteria:

* previous orthodontic treatment
* Probing depth values exceeding 3 mm
* Radiographic evidence of bone loss
* Regular administration medication that affects bone metabolism such as prolonged use of corticosteroids, or bisphosphonates and NSAIDs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Speed of tooth movement | Baseline (T1), post-treatment at time of debonding (T2), and 9 months post-treatment (T3).
  The total duration of active orthodontic treatment will be estimated in weeks from the time of starting the active orthodontic treatment, immediately following the corticotomy procedure, to the time of debonding.

SECONDARY OUTCOMES:
Bone density | Baseline (T1), post-treatment at time of debonding (T2), and 9 months post-treatment (T3).
  Bone density will be evaluated radiographically
Root length | Baseline (T1), post-treatment at time of debonding (T2), and 9 months post-treatment (T3).
  Root length will be evaluated radiographically

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdelaziz University. Faculty of dentistry, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bahammam MA. Effectiveness of bovine-derived xenograft versus bioactive glass with periodontally accelerated osteogenic orthodontics in adults: a randomized, controlled clinical trial. BMC Oral Health. 2016 Nov 30;16(1):126. doi: 10.1186/s12903-016-0321-x. PMID 27903250